CLINICAL TRIAL: NCT00002587
Title: A PHASE I STUDY OF PROLONGED LOW-DOSE TOPOTECAN INFUSION COMBINED WITH PACLITAXEL (TAXOL)
Brief Title: Paclitaxel Plus Topotecan in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02235; NYU-9315; NCI-T93-0115D; CDR0000063738 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-11 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2001-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Paclitaxel; Topotecan

ARMS (1):
- Arm I (Experimental): Patients receive paclitaxel IV over 3 hours on day 1 followed 2-6 hours later by topotecan IV continuously on days 1-14. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of topotecan and paclitaxel until the maximum tolerated dose (MTD) of each drug is determined. The MTD is defined as the highest dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: paclitaxel; Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
Phase I trial to study the effectiveness of paclitaxel plus topotecan in treating patients who have solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and quantitative and qualitative toxic effects of topotecan and paclitaxel in patients with solid tumors.

II. Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose escalation study of topotecan and paclitaxel.

Patients receive paclitaxel IV over 3 hours on day 1 followed 2-6 hours later by topotecan IV continuously on days 1-14. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan and paclitaxel until the maximum tolerated dose (MTD) of each drug is determined. The MTD is defined as the highest dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 10-20 patients will be accrued for this study within 8-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven solid tumor
* Measurable or evaluable disease
* Measurable disease defined as tumor outside prior radiotherapy fields and reproducibly measurable in 2 dimensions on physical exam, x-ray, CT, or MRI

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: 0 or 1
* Life expectancy: At least 12 weeks
* WBC at least 4,000/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.5 mg/dL
* AST less than 3 times normal
* Alkaline phosphatase less than 3 times normal
* Creatinine no greater than 1.5 mg/dL
* No poorly controlled angina
* No history of congestive heart failure
* No myocardial infarction within the past 6 months
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* No concurrent prophylactic hematopoietic growth factors
* No concurrent medications altering cardiac conduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1994-09; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States